CLINICAL TRIAL: NCT01948310
Title: Effects of Ranolazine and Exercise on Daily Physical Activity Trial
Acronym: EREDA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00045794
Record Dates: First submitted 2013-09-17; First posted 2013-09-23 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Chronic Stable Angina
MeSH Terms: conditions — Angina, Stable | interventions — Ranolazine; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranolazine plus Exercise (Active Comparator): Ranolazine 1000mg pill twice per day plus aerobic exercise three times per week, 45 minutes per session at an intensity of 10-20 beats per minute below the angina threshold.
  Interventions: Drug: Ranolazine; Behavioral: Aerobic Exercise
- Placebo plus Exercise (Placebo Comparator): Placebo pill twice per day plus aerobic exercise three times per week, 45 minutes per session at an intensity of 10-20 beats per minute below the angina threshold.
  Interventions: Behavioral: Aerobic Exercise; Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Comparison of Ranolazine 1000mg twice per day versus placebo twice per day
  Other Names: Renexa
  Arms: Ranolazine plus Exercise
Behavioral: Aerobic Exercise — Aerobic exercise 3 times per week, 45 minutes per session at an intensity of 10-20 beats per minute below the angina threshold (heart rate at which angina symptoms began on the stress test)
Drug: Placebo — Comparison of placebo twice per day vs. Ranolazine 1000mg twice per day
  Arms: Placebo plus Exercise

SUMMARY:
The primary objective is to assess whether the increased angina threshold on ranolazine and subsequent higher training intensity will result in improved exercise tolerance and oxygen consumption; and greater than that observed with exercise training on placebo. The study team anticipates the chronic exercise improvements with ranolazine will be incrementally higher than the acute effects provided by ranolazine alone and demonstrated in previous trials. Key secondary objectives include the acute ranolazine and chronic exercise plus ranolazine effects on total daily energy expenditure (TDEE) and angina-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Documented CAD diagnosis
* Stable angina ≥ 3 months

Exclusion Criteria:

* Class III or IV heart failure
* Myocardial Infarction or coronary revascularization procedure within 2 months
* QT interval > 500ms or prescribed medication known to prolong the QTc interval
* Contraindicated Medications
* Metformin dose > 1700mg/day
* Class Ia, Ic and III anti-arrhythmics
* CYP3A inhibitors
* Simvastatin >20mg/day
* Severe renal disease (< 30ml/min creatinine clearance)
* Currently on dialysis
* Lack of transportation to the exercise and testing facilities
* Implanted pacemaker that is not rate responsive

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-12; Primary Completion 2016-10-10 (Actual); Study Completion 2016-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William E Kraus, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Living, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-eight subjects were recruited for this study. One dropped out before randomization.
Period: Overall Study
Arm/Group | Placebo Plus Exercise | Ranolazine Plus Exercise
Started | 19 | 18
Completed | 16 | 13
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Plus Exercise | Ranolazine Plus Exercise | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (8.3) | 67.4 (11.2) | 68.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Oxygen Consumption (VO2 Max)
Description: This test involves exercising on a treadmill or bike to maximal exertion, during which the subject's breathing and oxygen consumption are measured. Under a set study protocol, treadmill or bike workload will increase every minute until the participant either chooses to end the test or the study personnel choose to end the test for safety purposes.
Time Frame: Baseline, Week 2 and Week 14
Population: Subjects who completed the study were included in the analysis
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Placebo Plus Exercise | Ranolazine Plus Exercise
Number analyzed (Participants) | 16 | 13
ml/kg/min
  Change at 2 weeks | 0.03 (1.2) | 0.38 (1.9)
  Change at 14 weeks | 0.9 (1.5) | 2.1 (3.4)
Statistical Analysis 1: Comparison: Placebo Plus Exercise; 2-0 weeks; Test type: Superiority; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo Plus Exercise; 0-14 weeks; Test type: Superiority; p = 0.03, t-test, 2 sided
Statistical Analysis 3: Comparison: Ranolazine Plus Exercise; 2-0 weeks; Test type: Superiority; p > 0.05, t-test, 2 sided
Statistical Analysis 4: Comparison: Ranolazine Plus Exercise; 14-0 weeks; Test type: Superiority; p = 0.005, t-test, 2 sided

2. Secondary Outcome: Change in Treatment Satisfaction as Measured by the Seattle Angina Questionnaire
Description: The Treatment Satisfaction scale is one of five scales of the Seattle Angina Questionnaire. The possible range of scores is 0 to 100, with higher scores indicating better quality of life.
Time Frame: Baseline, Week 2 and Week 14
Population: Subjects who completed the study were included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Plus Exercise | Ranolazine Plus Exercise
Number analyzed (Participants) | 16 | 13
units on a scale
  2-0 Weeks | 0.8 (9.1) | 5.3 (8.0)
  14-0 weeks | 3.1 (13.3) | -1.0 (13.0)
Statistical Analysis 1: Comparison: Placebo Plus Exercise; 2-0 weeks; Test type: Superiority; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo Plus Exercise; 14-0 weeks; Test type: Superiority; p > 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: Ranolazine Plus Exercise; 2-0 weeks; Test type: Superiority; p = 0.03, t-test, 2 sided
Statistical Analysis 4: Comparison: Ranolazine Plus Exercise; 14-0 weeks; Test type: Superiority; p > 0.05, t-test, 2 sided

3. Secondary Outcome: Change in Total Daily Energy Expenditure
Description: Total daily physical activity is measured via Actigraph GT3X accelerometers. Accelerometers will be worn for 7 days pre-drug, post-drug/pre-exercise (week 4) and again in the final month of the exercise intervention (week 13)
Time Frame: Week 1, Week 4 and Week 14
Population: Subjects who completed the study were included in the analysis.
Measure: Mean (Standard Deviation); unit: kj/hr
Arm/Group | Placebo Plus Exercise | Ranolazine Plus Exercise
Number analyzed (Participants) | 16 | 13
kj/hr
  2-0 weeks | 2.0 (39.3) | -7.6 (29.3)
  14-0 weeks | 22.2 (54.2) | 24.3 (29.9)
Statistical Analysis 1: Comparison: Placebo Plus Exercise; 2-0 weeks; Test type: Superiority; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo Plus Exercise; 0-14 weeks; Test type: Superiority; p = 0.13, t-test, 2 sided
Statistical Analysis 3: Comparison: Ranolazine Plus Exercise; 2-0 weeks; Test type: Superiority; p > 0.05, t-test, 2 sided
Statistical Analysis 4: Comparison: Ranolazine Plus Exercise; 14-0 weeks; Test type: Superiority; p = 0.013, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline until Week 14.
Arm/Group | Ranolazine Plus Exercise | Placebo Plus Exercise
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/18 | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine Plus Exercise (N=18) | Placebo Plus Exercise (N=19)
mild myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No